CLINICAL TRIAL: NCT06194656
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of SIBP-03 Injection Combined With Cetuximab in Patients With Recurrent/Metastatic Advanced Head and Neck Squamous Cell Carcinoma (Non-nasopharyngeal Carcinoma)
Brief Title: Clinical Trial of SIBP-03 in Patients With Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIBP-03-02
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck squamous cell carcinoma; safety; tolerability; pharmacokinetics; efficacy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: Ⅱa is an open-label study and Ⅱb is a randomized, double-blind study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): Experimental group in Ⅱa (part one). It will be the dose A of SIBP-03. It will determine whether the dose A is the optimal recommended dosage (RP2D) based on actual study results.
  Interventions: Drug: HER3 Monoclonal antibodies-Dose A; Combination Product: Cetuximab injection
- Group B (Experimental): Experimental group in Ⅱa (part one). It will be the dose B of SIBP-03. It will determine whether the dose B is the RP2D based on actual study results.
  Interventions: Drug: HER3 Monoclonal antibodies-Dose B; Combination Product: Cetuximab injection
- Group C (Experimental): Experimental group in Ⅱa (part two). It will be the dose C of SIBP-03. It will determine whether the dose C is the RP2D based on actual study results.
  Interventions: Drug: HER3 Monoclonal antibodies-Dose C; Combination Product: Cetuximab injection
- Group D (Experimental): Experimental group in Ⅱb. It will be the RP2D of SIBP-03.
  Interventions: Other: HER3 Monoclonal antibodies-Dose D; Combination Product: Cetuximab injection
- Group E (Placebo Comparator): Placebo of SIBP-03 (SIBP-03 solvent without HER3 antibody), and the dose will be the same with group D.
  Interventions: Other: Placebo; Combination Product: Cetuximab injection

INTERVENTIONS:
Drug: HER3 Monoclonal antibodies-Dose A — Dose A, intravenous infusion (IV), once every three weeks, 21 days as a cycle. The infusion time is 90 min (± 5 min).
  Arms: Group A
Drug: HER3 Monoclonal antibodies-Dose B — Dose B, intravenous infusion (IV), once every three weeks, 21 days as a cycle. The infusion time is 90 min (± 5 min).
  Arms: Group B
Drug: HER3 Monoclonal antibodies-Dose C — Dose C, intravenous infusion (IV), once every three weeks, 21 days as a cycle. The infusion time is 90 min (± 5 min).
  Arms: Group C
Other: HER3 Monoclonal antibodies-Dose D — The optimal recommended dosage (RP2D) of SIBP-03intravenous, infusion (IV), once every three weeks, 21 days as a cycle. The infusion time is 90 min (± 5 min).
  Arms: Group D
Other: Placebo — SIBP-03 solvent without HER3 antibody, intravenous infusion (IV), once every one weeks, 21 days as a cycle.
  Arms: Group E
Combination Product: Cetuximab injection — Medications used for combination therapy, intravenous infusion (IV). Administer once a week.

SUMMARY:
This phase II study will be conducted in two parts (Ⅱa and Ⅱb), with a 21-day treatment cycle until disease progression, intolerable toxicity, withdrawal of informed consent, death, initiation of new anti-tumor treatment or loss of follow-up.

DETAILED DESCRIPTION:
This phase II study will be conducted in two parts (Ⅱa and Ⅱb), with a 21-day treatment cycle until disease progression, intolerable toxicity, withdrawal of informed consent, death, initiation of new anti-tumor treatment or loss of follow-up. The participants in both study parts are the same, both of whom were patients with recurrent/metastatic advanced HNSCC (non nasopharyngeal carcinoma).

* a is an open-label study. Part one, 12 subjects were randomly assigned 1:1 to two groups and treated with SIBP-03 dose A or dose B every 3 weeks (Q3W) combined with cetuximab every week (QW). Part two, 3 subjects were treated with SIBP-03 dose C Q3W combined with cetuximab QW. If 1/3 subjects (1 case) have DLT, 3 more subjects need to continue to observe the safety and tolerance; If DLT occurs in 3 cases or ≥ 2 cases in 6 cases, the sponsor and the researcher will discuss and decide whether to terminate this part of the study or change the dose. 12 subjects were added at most.
* b is a randomized, double-blind study. Including an experimental group (RP2D) and a placebo control group. The qualified subjects in this stage will be randomly assigned according to the ratio of 2: 1, including 38 cases in the experimental group and 19 cases in the control group, with a total of 57 subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in the study and signed the informed consent.
* Male and female aged between 18 and 75 years old, regardless of gender.
* Patients with recurrent/metastatic advanced HNSCC who have been diagnosed by histology or cytology, progressed or intolerant after previous immunotherapy containing anti-PD-1/anti-PD-L1 and platinum, and have no indication of radical local treatment. Subjects should not receive more than 2 lines of treatment in the past.
* During the screening period, subjects must provide tumor tissues and blood samples for biomarker detection. If the subject does not have an archived tumor tissue sample, he or she will undergo a fresh tumor biopsy during the screening period to obtain the corresponding tumor sample. If the subject can't provide archived or fresh tumor tissue samples, but can provide the previous test reports of qualified institutions, including all biomarker indicators specified in this scheme, they can be screened after communicating with the sponsor.
* There must be at least one measurable lesion as the target lesion (according to RECIST v1.1 standard). Tumor lesions located in previous radiotherapy areas or other local regional treatment sites are generally not measurable lesions unless the lesion has definite progression.
* The ECOG physical fitness score is 0-1.
* The laboratory test results meet the requirements.
* The expected survival time is ≥ 3 months.
* In fertile female subjects, the blood pregnancy test must be negative within 7 days before the first medication. Subjects of reproductive age (including male subjects) had no family planning during the trial period and within 6 months after the last administration and voluntarily took effective contraceptive measures.

Exclusion Criteria:

* The primary site of squamous cell carcinoma is nasal cavity, paranasal sinuses, nasopharynx and salivary gland.
* The participant has received any HER3 targeting or EGFR targeting therapy in the past.
* Active central nervous system metastasis and/or meningeal metastasis.
* Previous allergy to human normal immunoglobulin or antibody preparation or other serious infusion reaction; Severe hypersensitivity disease, allergic constitution.
* In the past 5 years, the subjects had suffered from malignant tumors other than those treated in this study (except cured thyroid cancer, skin basal cell carcinoma and cervical carcinoma in situ).
* People infected with active human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B vrius (HBV), syphilis or active tuberculosis, and asymptomatic chronic hepatitis B or hepatitis C carriers may be excluded.
* The subjects have not recovered from the toxicity of previous anti-tumor therapy to grade ≤ 1 or baseline level (except participants with hair loss, neuropathy of grade ≤ 2 or stabilized thyroid function's decline by hormon replacement therapy).
* Subjects are currently participating in and receiving research treatment or have been treated with other research drugs or medical devices within 4 weeks before the first use of research drugs.
* Patients who plan to receive any other anti-tumor treatment during the trial should be excluded.
* Major surgery, radiotherapy (except palliative radiotherapy for targeted bone metastasis), or treatment such as unhealed surgical wound, ulcer or fracture within 4 weeks before the first administration; Received Chinese patent medicines or Chinese herbal medicines with anti-tumor indications within 2 weeks before the first administration; Chemotherapy was received within 3 weeks before the first administration, and anti-tumor treatments such as biotherapy, endocrine therapy, targeted therapy and immunotherapy were received within 4 weeks
* Those who have been vaccinated live within 30 days before the first administration.
* Active infections requiring systemic treatment, such as pneumonia, bacteremia, septicemia, etc.
* A history of pulmonary interstitial disease, pulmonary interstitial fibrosis or drug-induced interstitial pneumonia or other clinically serious lung diseases (CTCAE 5.0 grade III-IV).
* Pulmonary thromboembolism, arterial thrombosis and deep vein thrombosis formation (DVT) occurred within 6 months before screening, except for infusion set-related thrombosis.
* Have a history or evidence of cardiovascular (CV) risk.
* During the screening period, 12-lead electrocardiogram (ECG) measurement was performed in the research center (the average value of QTcF that needs to be measured repeatedly for 3 times), and the QT interval (QTcF) corrected by Fridericia method was > 450 milliseconds (male) or (QTcF) > 470 milliseconds (female); LVEF of cardiac ultrasound was less than 50%.
* Therapeutic surgery was performed within 28 days before the first administration, or major surgery was expected during the study period (except diagnosis, biopsy and drainage).
* People with mental disorders or poor compliance.
* Pregnant or lactating women.
* According to the researcher's judgment, there are accompanying diseases (such as severe hypertension, diabetes, thyroid diseases, etc.) that seriously endanger the patient's safety or affect the patient's completion of the study.
* Suffering from diseases requiring long-term treatment with high doses (defined as 30mg/d hydrocortisone or equivalent doses of other hormonal drugs) of hormones or immunosuppressive drugs.
* After active treatment, uncontrollable pleural and abdominal cavity or other lacunar effusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The occurrence of any adverse events (AE) | 30 days after the last dose
  All subjects after receiving the investigational drug were observed during the trial for any AE that occurred during the clinical study.AE were manifested as symptoms, signs, diseases, or abnormal laboratory tests, but may not necessarily have a causal relationship with the investigational drug.
SAE (Serious Adverse Events) | 30 days after the last dose
  That is serious adverse events, any serious adverse events that occurred to the subject during the study period.
Cmax (Peak Plasma Concentration) | 30 days after the last dose
  It shows the highest plasma concentration of a drug that can be achieved after administration.
Tmax(Peak Time) | 30 days after the last dose
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the subject plasma concentration curve after administration.
T ½(Terminal elimination half-life) | 30 days after the last dose
  It reflects how quickly the drug is eliminated from the body.
CL(Clearance Rate) | 30 days after the last dose
  Apparent volume of drug distribution removed from the body per unit time.
Difference of ORR | The 1 day the test results reported after the last dose
  Differences in ORR between SIBP-03 and placebo evaluated by the Independent Evaluation Committee (IRC) according to RECIST 1.1. Only applicable to part two.

SECONDARY OUTCOMES:
ORR (Objective Response Rate) | The 1 day the test results reported after the last dose
  The proportion of subjects whose tumor volume shrinks to a predetermined value and maintains the minimum time limit, and is the sum of complete and partial responses.
DCR (Disease control rate) | The 1 day the test results reported after the last dose
  In clinical trials, the percentage of subjects with advanced or metastatic cancer who responded fully to cancer treatment, partially responded, and had stable disease.
PFS (Progression-free survival) | The 1 day the test results reported after the last dose
  The time between the onset of randomization and the onset (of any aspect) of tumor progression or death (from any cause).
ADA (Anti-drug Antibody) | The 1 day the test results reported after the last dose
  The incidence of anti-drug antibody.
NAb (Neutralizing Antibody) | The 1 day the test results reported after the last dose
  The incidence of neutralizing antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Doctor, Principal Investigator — Shanghai Oriental Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No